CLINICAL TRIAL: NCT06748976
Title: EEG Alpha Rhythm Modulation Using Sham Neurofeedback During Attentional Control in a Virtual Reality Environment
Brief Title: Modulation of Cortical Brain Activity During Attentional Control
Status: Recruiting | Type: Observational
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, José Biurrun Manresa, Principal Investigator, National Council of Scientific and Technical Research, Argentina
Other Study IDs: IS004817
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Rumination; Chronic Pain; Fibromyalgia
Keywords: operant conditioning; rumination; metacognition; neurofeedback; selective attention
MeSH Terms: conditions — Rumination Syndrome; Chronic Pain; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy: Volunteers: Adults aged 18-60 years with normal or corrected vision, no clinical history of photosensitive epilepsy, psychiatric disorders, significant hearing loss, migraines, or substance abuse.
  Interventions:
  Positive sham-neurofeedback Negative sham-neurofeedback Control (no feedback)
  Interventions: Other: Positive sham neurofeedback; Other: Negative sham neurofeedback; Other: Control

INTERVENTIONS:
Other: Positive sham neurofeedback — Participants receive simulated positive reinforcement feedback designed to mimic successful modulation of EEG alpha rhythms, despite the feedback not being directly based on their actual neural activity. This condition aims to create the perception of improved attentional control.
Other: Negative sham neurofeedback — Participants receive simulated negative reinforcement feedback that mimics unsuccessful modulation of EEG alpha rhythms, regardless of their actual neural activity. This condition is intended to simulate reduced attentional control.
Other: Control — Participants perform the same attentional task but without receiving any feedback. This condition serves as a baseline to evaluate the effects of the sham neurofeedback interventions on EEG alpha rhythm modulation.

SUMMARY:
The goal of this study is to determine whether an open-loop sham neurofeedback system can effectively modulate EEG alpha rhythms, which are associated with attentional control. The main questions it aims to answer are:

Does positive sham neurofeedback lead to a decrease in relative EEG alpha power compared to a control condition without feedback?

Researchers will compare the effects of positive and negative sham-neurofeedback conditions to a control condition without feedback to assess the system's impact on alpha rhythm modulation. Participants will:

Experience three conditions (positive sham-neurofeedback, negative sham-neurofeedback, and no feedback) within a virtual reality environment.

Undergo EEG recordings to measure changes in alpha power as a marker of attentional resource allocation.

Provide written informed consent and complete the study following ethical guidelines.

This study seeks to explore the potential of open-loop feedback systems to enhance attentional control by modulating alpha rhythm.

DETAILED DESCRIPTION:
Attention is a vital cognitive process that enables selective focus on behaviourally relevant information. A perceived lack of attentional control has been linked to mental disorders such as depression and anxiety, often manifesting through maladaptive coping strategies like rumination. As a trainable cognitive skill, attentional control can be enhanced through learning processes, particularly when reinforced by positive feedback within a classical operant conditioning framework. EEG studies have demonstrated that decreases in alpha rhythm power are associated with increased attentional resource allocation. While neurofeedback systems, especially those targeting alpha rhythms, typically rely on closed-loop modulation during attentional tasks, the impact of open-loop feedback on EEG alpha modulation remains unexplored. This study aims to determine whether an open-loop feedback system can effectively modulate EEG alpha rhythms, as a marker correlate of attentional control. The investigators propose a within-subject experiment where participants will experience positive and negative sham neurofeedback conditions, as well as a control condition with no feedback, all within a virtual reality environment. The investigators hypothesize that relative EEG alpha power will decrease in the positive sham neurofeedback condition compared to the control condition, reflecting a meaningful increase in attentional resource allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 60 years.
* Normal or corrected vision.
* Ability to provide written informed consent.

Exclusion Criteria:

* Diagnosed with photosensitive epilepsy.
* Significant hearing loss or diagnosed hearing impairment.
* Current psychiatric illness or disorder.
* History of migraines or chronic headaches.
* History of substance or alcohol abuse.
* Currently pregnant.
* Discomfort with using a virtual reality headset, assessed during a pilot session.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include adults aged between 18 and 60 years, selected from the city of Paraná and surrounding areas. The population will be balanced in terms of age and gender, ensuring representation across two age groups (18-40 years and 41-60 years).
  Participants will be recruited through:
  * Word-of-mouth.
  * Social media platforms.
  * University mailing lists and community boards. Initial contact will be made via telephone or email, where potential participants will be provided with detailed information about the study's purpose, procedures, and eligibility criteria. Recruitment materials and communications will describe the study as a conventional neurofeedback experiment to maintain participant naivety about the specific hypotheses and experimental conditions.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Relative alpha power | Immediately after intervention
  The primary outcome of the study is the change in relative EEG alpha power during the positive sham-neurofeedback condition compared to the control condition (no feedback). A decrease in relative alpha power is interpreted as an indicator of increased attentional resource allocation, reflecting enhanced attentional control. This measure is derived from EEG recordings captured during the experimental tasks in each condition.

SECONDARY OUTCOMES:
Relative alpha power | Immediately after intervention
  The secondary outcome of the study is the change in relative EEG alpha power during the negative sham-neurofeedback condition compared to the control condition (no feedback).

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Ingeniería, Universidad Nacional de Entre Ríos, Oro Verde, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available on the 'Open Science Framework' after undergoing the process of anonymization to remove any participant-identifying information. The data will consist of the raw EEG signals and raw behavioral responses. Additionally, the statistical analysis and Python notebooks used to process the data will also be shared
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The participant's data and the processing pipeline will be available after the data collection is finished. The supporting information (including the study protocol, the statistical analysis plan and the informed consent) will be uploaded as soon as possible.
Access Criteria: The data will be publicly available.

REFERENCES:
- [Background] Knowles MM, Wells A. Single Dose of the Attention Training Technique Increases Resting Alpha and Beta-Oscillations in Frontoparietal Brain Networks: A Randomized Controlled Comparison. Front Psychol. 2018 Sep 20;9:1768. doi: 10.3389/fpsyg.2018.01768. eCollection 2018. PMID 30294294
- [Background] Magosso E, Ricci G, Ursino M. Modulation of brain alpha rhythm and heart rate variability by attention-related mechanisms. AIMS Neurosci. 2019 Mar 4;6(1):1-24. doi: 10.3934/Neuroscience.2019.1.1. eCollection 2019. PMID 32341965
- [Background] Enriquez-Geppert S, Smit D, Pimenta MG, Arns M. Neurofeedback as a Treatment Intervention in ADHD: Current Evidence and Practice. Curr Psychiatry Rep. 2019 May 28;21(6):46. doi: 10.1007/s11920-019-1021-4. PMID 31139966